CLINICAL TRIAL: NCT03948880
Title: Incidence of OIRD in Medical and Trauma Patients on the General Care Floor Receiving PCA or Nurse Administered Intravenous Opioids Monitored by Capnography and Pulse Oximetry: A Prospective, Blinded Observational Study
Brief Title: Incidence OIRD Medical and Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fresno Community Hospital and Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Susan Dempsey Ortega, Clinical Nurse Specialist, Fresno Community Hospital and Medical Center
Other Study IDs: FresnoCHMC
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Depression; Sedation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this prospective, blinded observational study is to correlate assessment of sedation and respiratory status with capnography and pulse oximetry monitoring in hospitalized adult medical and trauma patients receiving patient-controlled analgesia (PCA) or nurse administered intravenous opioids for acute pain. Nursing assessment of respiratory status and sedation level will be correlated with capnography and pulse oximetry values as technology-supported monitoring to identify respiratory depression and opioid-induced sedation. The secondary objective is to identify capnography and pulse oximetry values that correlate with respiratory decompensation and opioid-induced sedation in medical and trauma patients on the general care floor.

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneously breathing adults 18 to 89 years of age
2. Receiving PCA or nurse administered IV opioids for medical or trauma-related pain
3. Admitted to the general care floor from the emergency department
4. Able to provide written informed consent

Exclusion Criteria:

1. Age is less than 18 years or greater than 89 years
2. Transfer to the general care floor from the ICU
3. Provider order for respiratory monitoring using continuous capnography
4. Receiving intrathecal or epidural opioids
5. Trauma patient with a nerve block
6. Inability or unwillingness to wear the EtCO2 sampling line nasal cannula or pulse oximetry sensor
7. History or diagnosis of a sleep disordered breathing syndrome
8. Use of CPAP or BIPAP non-invasive ventilation as home regime
9. Pre-existing co-morbidity that impacts respiration or ventilation (e.g. COPD or pulmonary fibrosis) (for the purpose of this study a trauma patient with rib fractures is not considered having a pre-existing condition)
10. Receiving non-invasive ventilation
11. Unable or unwilling to participate
12. Member of a vulnerable population such as pregnant women or prisoners

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will be hospitalized, adult medical or trauma patients on the general care floor receiving patient-controlled analgesia or nurse administered intravenous opioids for acute pain.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2019-10-29 (Estimated); Study Completion 2019-11-29 (Estimated)

PRIMARY OUTCOMES:
Hypoventilation | Change from baseline measurement observed within 60 minutes after opioid administration
  The number of subjects who experience hypoventilation using respiratory monitoring with continuous capnography for data collection.
Hypoventilation | Change from baseline measurement observed within 60 minutes after opioid administration
  The percentage of subjects who experience hypoventilation using respiratory monitoring with continuous capnography for data collection.
Hypoventilation | Change from baseline measurement observed within 60 minutes after opioid administration
  The characteristics of subjects who experience hypoventilation using respiratory monitoring with continuous capnography for data collection.

SECONDARY OUTCOMES:
Hypoxemia | Change from baseline measurement observed within 60 minutes after opioid administration ]
  The number of subjects who experience oxygen desaturation using respiratory monitoring with continuous pulse oximetry for data collection.
Hypoxemia | Change from baseline measurement observed within 60 minutes after opioid administration ]
  The percentage of subjects who experience oxygen desaturation using respiratory monitoring with continuous pulse oximetry for data collection.
Hypoxemia | Change from baseline measurement observed within 60 minutes after opioid administration ]
  The characteristics of subjects who experience oxygen desaturation using respiratory monitoring with continuous pulse oximetry for data collection.

OTHER OUTCOMES:
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration ]
  The number of subjects who experience unintended sedation using the Pasero Opioid-Induced Sedation Scale in which sedation levels of S, 1, 2, 3, 4 are assessed where "S" represents normal sleep, increasing numbers represent increasing levels of sedation, and sedation levels 3 or 4 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration ]
  The percentage of subjects who experience unintended sedation using the Pasero Opioid-Induced Sedation Scale in which sedation levels of S, 1, 2, 3, 4 are assessed where "S" represents normal sleep, increasing numbers represent increasing levels of sedation, and sedation levels 3 or 4 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration ]
  The characteristics of subjects who experience unintended sedation using the Pasero Opioid-Induced Sedation Scale in which sedation levels of S, 1, 2, 3, 4 are assessed where "S" represents normal sleep, increasing numbers represent increasing levels of sedation, and sedation levels 3 or 4 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The number of subjects who experience unintended sedation using the Moline Roberts Pharmacologic Sedation Scale in which sedation levels of 1, 2, 3, 4, 5, 6 are assessed where increasing numbers represent increasing levels of sedation and sedation levels 3 or 4 or 5 or 6 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The percentage of subjects who experience unintended sedation using the Moline Roberts Pharmacologic Sedation Scale in which sedation levels of 1, 2, 3, 4, 5, 6 are assessed where increasing numbers represent increasing levels of sedation and sedation levels 3 or 4 or 5 or 6 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The characteristics of subjects who experience unintended sedation using the Moline Roberts Pharmacologic Sedation Scale in which sedation levels of 1, 2, 3, 4, 5, 6 are assessed where increasing numbers represent increasing levels of sedation and sedation levels 3 or 4 or 5 or 6 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The number of subjects who experience unintended sedation using the Richmond Agitation Sedation Scale in which sedation levels of +4, +3, +2, +1, 0, -1, -2, -3, -4, -6 are assessed where decreasing numbers represent increasing levels of sedation and sedation levels of -1 or -2 or -3 or -4 or -5 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The percentage of subjects who experience unintended sedation using the Richmond Agitation Sedation Scale in which sedation levels of +4, +3, +2, +1, 0, -1, -2, -3, -4, -6 are assessed where decreasing numbers represent increasing levels of sedation and sedation levels of -1 or -2 or -3 or -4 or -5 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  The characteristics of subjects who experience unintended sedation using the Richmond Agitation Sedation Scale in which sedation levels of +4, +3, +2, +1, 0, -1, -2, -3, -4, -6 are assessed where decreasing numbers represent increasing levels of sedation and sedation levels of -1 or -2 or -3 or -4 or -5 indicate unintended opioid-induced sedation for the purpose of this study

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Dempsey, PhD(c), Principal Investigator — UCLA and Community Regional Medical Center
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen LW, Berg KM, Chase M, Cocchi MN, Massaro J, Donnino MW; American Heart Association's Get With The Guidelines((R))-Resuscitation Investigators. Acute respiratory compromise on inpatient wards in the United States: Incidence, outcomes, and factors associated with in-hospital mortality. Resuscitation. 2016 Aug;105:123-9. doi: 10.1016/j.resuscitation.2016.05.014. Epub 2016 May 30. PMID 27255952
- [Background] Arozullah AM, Khuri SF, Henderson WG, Daley J; Participants in the National Veterans Affairs Surgical Quality Improvement Program. Development and validation of a multifactorial risk index for predicting postoperative pneumonia after major noncardiac surgery. Ann Intern Med. 2001 Nov 20;135(10):847-57. doi: 10.7326/0003-4819-135-10-200111200-00005. PMID 11712875
- [Background] Belcher AW, Khanna AK, Leung S, Naylor AJ, Hutcherson MT, Nguyen BM, Makarova N, Sessler DI, Devereaux PJ, Saager L. Long-Acting Patient-Controlled Opioids Are Not Associated With More Postoperative Hypoxemia Than Short-Acting Patient-Controlled Opioids After Noncardiac Surgery: A Cohort Analysis. Anesth Analg. 2016 Dec;123(6):1471-1479. doi: 10.1213/ANE.0000000000001534. PMID 27607476
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Canet J, Sabate S, Mazo V, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P; PERISCOPE group. Development and validation of a score to predict postoperative respiratory failure in a multicentre European cohort: A prospective, observational study. Eur J Anaesthesiol. 2015 Jul;32(7):458-70. doi: 10.1097/EJA.0000000000000223. PMID 26020123
- [Background] Cashman JN, Dolin SJ. Respiratory and haemodynamic effects of acute postoperative pain management: evidence from published data. Br J Anaesth. 2004 Aug;93(2):212-23. doi: 10.1093/bja/aeh180. Epub 2004 May 28. PMID 15169738
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Dahan A, Aarts L, Smith TW. Incidence, Reversal, and Prevention of Opioid-induced Respiratory Depression. Anesthesiology. 2010 Jan;112(1):226-38. doi: 10.1097/ALN.0b013e3181c38c25. PMID 20010421
- [Background] Dempsey, SF, Khanna, AK, Buhre, W, Saager, L, DiStefano, P, Weingarten, T., Dahan, A., Brazzi, L., Overdyk, F., McIntyre, R. Incidence of Respiratory Depression and Derivation of a Novel Opioid-Induced Respriatory Depression Risk Prediction Tool. Poster presentation. UCLA School of Nursing Research Day, May 14, 2019.
- [Background] Gupta K, Prasad A, Nagappa M, Wong J, Abrahamyan L, Chung FF. Risk factors for opioid-induced respiratory depression and failure to rescue: a review. Curr Opin Anaesthesiol. 2018 Feb;31(1):110-119. doi: 10.1097/ACO.0000000000000541. PMID 29120929
- [Background] Izrailtyan I, Qiu J, Overdyk FJ, Erslon M, Gan TJ. Risk factors for cardiopulmonary and respiratory arrest in medical and surgical hospital patients on opioid analgesics and sedatives. PLoS One. 2018 Mar 22;13(3):e0194553. doi: 10.1371/journal.pone.0194553. eCollection 2018. PMID 29566020
- [Background] Jarzyna D, Jungquist CR, Pasero C, Willens JS, Nisbet A, Oakes L, Dempsey SJ, Santangelo D, Polomano RC. American Society for Pain Management Nursing guidelines on monitoring for opioid-induced sedation and respiratory depression. Pain Manag Nurs. 2011 Sep;12(3):118-145.e10. doi: 10.1016/j.pmn.2011.06.008. PMID 21893302
- [Background] Khanna, A, Buhre, W, Saager, L, DiStefano, P, Weingarten, R, Dahan, A, Brazzi, L, & Overdyk, R. Derivation and validation of a novel opioid-induced respiratory depression risk predication tool. Critical Care Medicine 47(1):36, 2019.
- [Background] Khanna AK, Sessler DI, Sun Z, Naylor AJ, You J, Hesler BD, Kurz A, Devereaux PJ, Saager L. Using the STOP-BANG questionnaire to predict hypoxaemia in patients recovering from noncardiac surgery: a prospective cohort analysis. Br J Anaesth. 2016 May;116(5):632-40. doi: 10.1093/bja/aew029. PMID 27106966
- [Background] Kessler ER, Shah M, Gruschkus SK, Raju A. Cost and quality implications of opioid-based postsurgical pain control using administrative claims data from a large health system: opioid-related adverse events and their impact on clinical and economic outcomes. Pharmacotherapy. 2013 Apr;33(4):383-91. doi: 10.1002/phar.1223. PMID 23553809
- [Background] Lam T, Nagappa M, Wong J, Singh M, Wong D, Chung F. Continuous Pulse Oximetry and Capnography Monitoring for Postoperative Respiratory Depression and Adverse Events: A Systematic Review and Meta-analysis. Anesth Analg. 2017 Dec;125(6):2019-2029. doi: 10.1213/ANE.0000000000002557. PMID 29064874
- [Background] Lee LA, Caplan RA, Stephens LS, Posner KL, Terman GW, Voepel-Lewis T, Domino KB. Postoperative opioid-induced respiratory depression: a closed claims analysis. Anesthesiology. 2015 Mar;122(3):659-65. doi: 10.1097/ALN.0000000000000564. PMID 25536092
- [Background] Morrison LJ, Neumar RW, Zimmerman JL, Link MS, Newby LK, McMullan PW Jr, Hoek TV, Halverson CC, Doering L, Peberdy MA, Edelson DP; American Heart Association Emergency Cardiovascular Care Committee, Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on P. Strategies for improving survival after in-hospital cardiac arrest in the United States: 2013 consensus recommendations: a consensus statement from the American Heart Association. Circulation. 2013 Apr 9;127(14):1538-63. doi: 10.1161/CIR.0b013e31828b2770. Epub 2013 Mar 11. No abstract available. PMID 23479672
- [Background] Overdyk FJ, Dowling O, Marino J, Qiu J, Chien HL, Erslon M, Morrison N, Harrison B, Dahan A, Gan TJ. Association of Opioids and Sedatives with Increased Risk of In-Hospital Cardiopulmonary Arrest from an Administrative Database. PLoS One. 2016 Feb 25;11(2):e0150214. doi: 10.1371/journal.pone.0150214. eCollection 2016. PMID 26913753
- [Background] Perman SM, Stanton E, Soar J, Berg RA, Donnino MW, Mikkelsen ME, Edelson DP, Churpek MM, Yang L, Merchant RM; American Heart Association's Get With the Guidelines(R)-Resuscitation (formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Location of In-Hospital Cardiac Arrest in the United States-Variability in Event Rate and Outcomes. J Am Heart Assoc. 2016 Sep 29;5(10):e003638. doi: 10.1161/JAHA.116.003638. PMID 27688235
- [Background] Ronen M, Weissbrod R, Overdyk FJ, Ajizian S. Smart respiratory monitoring: clinical development and validation of the IPI (Integrated Pulmonary Index) algorithm. J Clin Monit Comput. 2017 Apr;31(2):435-442. doi: 10.1007/s10877-016-9851-7. Epub 2016 Mar 9. PMID 26961501
- [Background] Stites M, Surprise J, McNiel J, Northrop D, De Ruyter M. Continuous Capnography Reduces the Incidence of Opioid-Induced Respiratory Rescue by Hospital Rapid Resuscitation Team. J Patient Saf. 2021 Sep 1;17(6):e557-e561. doi: 10.1097/PTS.0000000000000408. PMID 28731933
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Background] Taenzer AH, Pyke JB, McGrath SP, Blike GT. Impact of pulse oximetry surveillance on rescue events and intensive care unit transfers: a before-and-after concurrence study. Anesthesiology. 2010 Feb;112(2):282-7. doi: 10.1097/ALN.0b013e3181ca7a9b. PMID 20098128
- [Background] Safe use of opioids in hospitals. Sentinel Event Alert. 2012 Aug 8;(49):1-5. No abstract available. PMID 22888503
- [Background] Weingarten TN, Herasevich V, McGlinch MC, Beatty NC, Christensen ED, Hannifan SK, Koenig AE, Klanke J, Zhu X, Gali B, Schroeder DR, Sprung J. Predictors of Delayed Postoperative Respiratory Depression Assessed from Naloxone Administration. Anesth Analg. 2015 Aug;121(2):422-9. doi: 10.1213/ANE.0000000000000792. PMID 25993390